CLINICAL TRIAL: NCT01308554
Title: Analgesic Efficacy of Ultrasound-guided Single Shot Subcostal Transversus Abdominis Plane (TAP) Block After Laparoscopic Gastric Bypass.
Brief Title: Pain Relieving Efficacy of TAP Block in Patients After Laparoscopic Gastric Bypass.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Funch-Jensen, Peter, M.D., D.M.Sc. (Individual)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TAP1
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Pain; Obesity; Surgery; Neuromuscular Inhibition
Keywords: TAP block; Pain; Obesity; Surgery; Laparoscopic gastric bypass
MeSH Terms: conditions — Pain; Obesity | interventions — Saline Waters; Saline Solution; Sodium Chloride; Salts; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sterile normal saline (Placebo Comparator): Control group will receive sterile normal saline in the block
  Interventions: Drug: Placebo: sterile normal saline
- Marcaine (Active Comparator): Study group will receive a bilateral TAP block using 20 ml of Marcaine 2,5 mg/ml on each side.
  Interventions: Drug: Marcaine

INTERVENTIONS:
Drug: Placebo: sterile normal saline — Bilateral TAP block using 20 ml of normal sterile saline per block.
  Other Names: Saline water; Saline solution; Sodium chloride; NaCl; Salt
  Arms: Sterile normal saline
Drug: Marcaine — Study group will receive a bilateral TAP block using 20 ml of 0,25% Marcain on each side.
  Other Names: Bupivacaine
  Arms: Marcaine

SUMMARY:
The purpose of this study is to determine whether injection of bupivacaine into the TAP is effective in the treatment of post operative pain after laparoscopic gastric bypass

DETAILED DESCRIPTION:
Obesity surgery is expensive, although highly competitive to the cost of obesity related disease. An important step would be to reorganize obesity surgery into a day surgical procedure. Some reports already exist in the literature but the number of publications are sparse, and the description of the condition of the patient is limited. Our primary aim, therefore, is to investigate the influence transverses abdominis plane block has on pain after laparoscopic gastric bypass.

The benefits of adequate postoperative analgesia are clear, and include a reduction in the postoperative stress response, reduction in postoperative morbidity and in certain types of surgery, improved surgical outcome. The benefits of utilizing regional analgesic techniques compared to systemic analgesics include reduction in pain intensity, decreased incidence of side effects from systemic analgesics and improved patient comfort. Effective pain control thereby accelerates recovery from surgery.

A substantial component of the pain experienced by patients after abdominal surgery is derived from the abdominal wall incision.

The Transversus Abdominis Plane (TAP) Block was first described in 2001 in a letter by Dr. Rafi. McDonnell et al have developed and tested the block and describes it as a landmark technique. TAP Block involves blocking the sensory afferent nerves that supply the anterior abdominal wall including the skin, muscles and the parietal peritoneum. Hebbard et al subsequently described an ultrasound guided technique for the TAP block which they named the Posterior TAP block. The posterior TAP block provides analgesia on the lower abdominal wall. Hebbard also described another ultrasound-guided technique called the Oblique Sub costal TAP block which provides analgesia for surgery on the upper abdominal wall.

There is some debate over the extent of sensory blockade achieved by TAP block. Nerves supplying the anterior abdominal wall are derived from T16 to L1 and pass through this plane before supplying the anterior abdominal wall. Earlier studies showed a T7-L1 spread of the block after a single posterior TAP injection, while some newer studies revealed that the block failed to spread above T10 so was suitable only for lower abdominal procedures. In contrast the oblique sub costal TAP block can provide an effective analgesia after surgery that involves dermatome T6 to T10, in other word provide analgesia for surgery on the upper abdominal wall.

Studies looking at posterior TAP block have demonstrated reduced postoperative morphine consumption and improved pain scores at rest and on movement in patients undergoing lower midline laparotomy, open appendectomy, laparoscopic appendectomy total abdominal hysterectomy, caesarean section and laparoscopic cholecystectomy. The duration of the morphine-sparing effect after a single shot injection into the posterior TAP has been reported to range from 12 to 48 hours. Pain scores both in rest and on movement are reduced compared to placebo in up to 48 hours after surgery. Single shot TAP blocks have also been used to provide analgesia in patients admitted to the ICU the analgesia provided by the block lasted between 16 to 24 hours.

There has been a report from Leicester General Hospital of the effectiveness of inserting catheters into the oblique sub costal TAP. The obtained block provided analgesia for more than 72 hours in patients who have had surgery on the upper abdominal wall (hepatobiliary surgery). They also describe the block as being effective rescue analgesia in patients in whom the epidural is ineffective.

Currently there are to our knowledge no clinical trials on the analgesic efficacy of single shot oblique sub costal TAP blocks for surgery of the upper abdominal wall. Niraj et al reports that they have observed the duration of postoperative analgesia to be 6 to 8 hours after single shot sub costal TAP. While Patil et al reports of sensory blockade for 5 hours along the dermatomal level T7-L1 after single shot posterior TAP block combined with sub costal TAP block.

Oblique sub costal TAP block could be a viable alternative for providing analgesia during the postoperative period. The block can be performed easily using ultrasound guidance, has an excellent safety profile, provides effective dynamic analgesia and has a significant morphine-sparing effect.

The proposed study involves the utilization of ultrasound to locate the oblique subcostal TAP, injection of bupivacaine or placebo (saline) into the TAP on each side and comparison of the analgesic efficacy of the TAP injection with that of placebo during two weeks in patients who have had gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged over 18 years who are scheduled for elective gastric bypass (incisions with the lower end of the incision at or above thoracic T 10 dermatome)

Exclusion Criteria:

* Lack of consent including from those patients who lack mental capacity to give informed consent
* Patients with history of drug allergy to bupivacaine
* Patients with history of chronic pain conditions: defined as patients with history of pain for above 3 months and who consume regular analgesics for their chronic pain
* American Society of Anesthesiologists (ASA) Class 4 and 5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
24h morphine consumption | 24h after the block is given

SECONDARY OUTCOMES:
Post operative nausea score | Before surgery and every second hour after surgery until nighttime and again three measurements each day for two weeks.
  none = 0; mild = 1; moderate = 2; severe = 3
Measurement of lung function (FEV1 and FVC) | Before surgery and 24h after.
The Verbal Analogue Scale (VAS) scores at rest and on moving | Before surgery and every second hour after surgery until nighttime and again three measurements each day for two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Funch-Jensen, D.M.Sc., Principal Investigator — Privathospital Hamlet Aarhus, Denmark
Locations (1):
- Privathospitalet Hamlet Aarhus, Aarhus N, Denmark